CLINICAL TRIAL: NCT07116083
Title: Diagnostic Performance of µQFR for Residual Functional Stenosis in Bifurcation Lesions After Single-stenting Strategy
Brief Title: µQFR for Branch Stenosis After Single Stent in Bifurcation Lesions
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Junbo Ge, Head of Department of Cardiology, Shanghai Zhongshan Hospital
Other Study IDs: ZSCD2025-01
Record Dates: First submitted 2025-07-28; First posted 2025-08-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Coronary Artery Disease (Left Main); Obstructive Coronary Artery Disease; Stent Implantation
Keywords: Functional Flow Reserve; Quantitative Flow Ratio
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main stent before branch balloon: Patiens is allocated pot-hoc to this group if the operator performs the single stent in the main branch first and follows with balloon expansion in the ostium of the side branch. Angiography will be saved anonymously and sent to an independent core lab for µQFR calculation. Operaters are blinded to µQFR results. µQFR measurement will be repeated before and after intervention in both main and side branches.
- Main stent after branch balloon: Patiens is allocated pot-hoc to this group if the operator performs expend the ostium of the side branch and then plants the single stent in the main branch. Angiography will be saved anonymously and sent to an independent core lab for µQFR calculation. Operaters are blinded to µQFR results. µQFR measurement will be repeated before and after intervention in both main and side branches.

SUMMARY:
Murray-law based single-view quantitative flow ratio (µQFR) has been recommended for guiding percutaneous coronary intervention (PCI) in selective patients. However, it's reliability has not been validated in bifurcation lesions which present complex anatomy and flluid conditions before and after PCI. The goal of this study is to investigate the diagnostic performance of µQFR in side branch after single-stent treatment for bifurcation lesions in patient with obstructive coronary artery diseases.

DETAILED DESCRIPTION:
The Murray law-based quantitative flow ratio (µQFR), derived from single-view angiography, is an established computational method for non-invasive functional assessment of coronary stenoses. Its utility in guiding percutaneous coronary intervention (PCI) in selected patients with straightforward lesions is recognized. However, its diagnostic reliability remains unvalidated in the context of coronary bifurcation lesions. These lesions exhibit inherent geometric and hemodynamic complexity due to altered flow patterns and shear stress distribution, both pre- and post-intervention. This complexity is particularly pertinent to side branches following single-stent strategies. Significant alterations in the local hemodynamic environment occur after stent deployment in the main vessel, potentially impacting side branch physiology and the accuracy of µQFR calculations specifically within this branch. Consequently, an evidence gap persists regarding the performance of µQFR for functional evaluation of the side branch after bifurcation PCI. This study specifically aims to evaluate the diagnostic performance of µQFR for assessing the functional significance of side branch stenoses after single-stent treatment of bifurcation lesions in patients with obstructive coronary artery disease (CAD). The primary objective is to determine the diagnostic performance of post-procedural µQFR measurements within the side branch of such complex lesions. The second objective is to investigate potential factors influencing the diagnostic performance of µQFR.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and provision of written informed consent for biospecimen donation upon hospital admission.
2. Clinical suspicion or diagnosis of CAD requiring coronary angiography and physiological assessment.
3. Angiographically confirmed true bifurcation lesions, including but not limited to: left main-left anterior descending-left circumflex (LM-LAD-LCx), left anterior descending-diagonal (LAD-Dg), left circumflex-obtuse marginal (LCx-OM), and right coronary artery-posterior left ventricular-posterior descending artery (RCA-PLV-PDA).
4. Bifurcation lesion vessel diameter ≥ 2.5 mm with visually estimated angiographic diameter stenosis ≥ 50%.

Exclusion Criteria:

1. Acute myocardial infarction.
2. Cardiogenic shock or severe heart failure (Killip class IV).
3. Serum creatinine > 150 μmol/L or estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73 m² calculated using the CKD-EPI formula.
4. Known allergy to iodinated contrast media.
5. History of coronary artery bypass graft surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with obstructive bifurcation lesions who intended to undergo single-stent treatment.
Sampling Method: Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of µQFR in side branch | Perioperative
  The diagnostic accuracy of µQFR in assessing ischemia in the side branch, using FFR as the gold standard, following main vessel stenting.

SECONDARY OUTCOMES:
Diagnostic accuracy of µQFR in main branch | Perioperative
  The effect of intravascular ultrasound (IVUS)-derived parameters on the diagnostic performance of µQFR in assessing ischemia in the main branch before and after stenting, using FFR as the gold standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
IPD sharing might be possible upon reasonable requirement and under institutional administrative regulations.